CLINICAL TRIAL: NCT03608332
Title: Diaphragmatic Ultrasound as a Guide Tool During Weaning From Mechanical Ventilation (Randomized Controlled Trial)
Brief Title: Diaphragmatic Ultrasound as a Guide Tool During Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DUS in weaning
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Diaphragmatic Ultrasound in Weaning

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (No Intervention): weaning readiness will be evaluated with the standard criteria :- A) Clinical assessment:-
  * Resolution of acute phase of disease for which patient was intubated
  * Adequate cough
  * Absence of excessive tracheobronchial secretions
  B) Objective criteria:-
  * Adequate oxygenation:PaO2>60mmHg with PEEP<8,SaO2>90%,FIO2 <0.5,PaO2/FIO2>200
  * Respiratory rate <30
  * PH and PaCO2 appropriate for patients' baseline respiratory status
  * Hemodynamically stable :minimal or no vasopressor/inotropes,no evidence of myocardial ischemia
  * HR<140 beats/minute
  * Patient is arousable or Glasgow coma scale (GCS)>13
- Group SD (Experimental): weaning readiness will be evaluated with the following criteria:- A) Clinical assessment:-
  * Resolution of acute phase of disease for which patient was intubated
  * Adequate cough
  * Absence of excessive tracheobronchial secretions
  B) Objective criteria:-
  * Adequate oxygenation:PaO2>60mmHg with PEEP<8,SaO2>90%,FIO2 <0.5,PaO2/FIO2>200
  * Respiratory rate <30
  * PH and PaCO2 appropriate for patients' baseline respiratory status
  * Hemodynamically stable :minimal or no vasopressor/inotropes,no evidence of myocardial ischemia
  * HR<140 beats/minute
  * Patient is arousable or Glasgow coma scale (GCS)>13
  C) Ultrasound criteria:-
  • Diaphragmatic excursion >11 mm
  Interventions: Device: diaphragmatic ultrasound

INTERVENTIONS:
Device: diaphragmatic ultrasound — Diaphragmatic excursion; Diaphragmatic movement will be measured with a 3.5-MHz US probe (Mindray machine, DC-N6).
  Arms: Group SD

SUMMARY:
To assess value of adding ultrasound derived variables to the usual parameters on success rate of weaning from mechanical ventilation in critically ill patients and to validate sensitivity and specificity of ultrasound derived variables (thickening fraction /diaphragmatic excursion)

DETAILED DESCRIPTION:
Difficult weaning from mechanical ventilation (MV) is a common problem in critically ill patients. Many parameters have been developed to aid weaning from MV such as P/F ratio (PO2/FiO2) and rapid shallow breathing index (respiratory rate/tidal volume), however, sensitivity and specificity for most variables are still variable in literature.

Multiple studies have found that patients tolerantof SBTs were found to have successful discontinuationsat least 77% of the time.

Causes of weaning failure include: airway and lung dysfunction, brain dysfunction, cardiac dysfunction, diaphragm dysfunction, and endocrine dysfunction .

Diaphragmatic dysfunction is a common cause of weaning failure , however most of the traditional methods used for evaluation of diaphragmatic function (fluoroscopy, trans-diaphragmatic pressure measurement) are invasive and not available.

Ultrasound assessment of diaphragmatic function has been developed recently providing an easy and safe method for evaluation of diaphragmatic excursion and thickening.

It was found that weaning failure (Re-intubation within 48 hours) was associated with diaphragmatic excursion <1 cm and thickening fraction <28% several studies reported the value of diaphragmatic ultrasound to predict weaning failure ,however no one of them used diaphragmatic ultrasound to guide weaning.

previous studies showed that failure rate of weaning from mechanical ventilation was 27% ,however failure rate in our department was 43% adding ultrasound derived values aims for improving success rate of weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients intubated for more than 48 hours who are ready for weaning

Exclusion Criteria:

* • Age < 18 years

  * surgical dressings over the right lower rib cage which would preclude ultrasound examination
  * patients with chest trauma, thoracotomy, diaphragmatic paralysis, diaphragmatic injury and diaphragmatic surgery
  * patients with neuromuscular diseases ( myasthenia gravis ,Muscular dystrophies ,Multiple sclerosis and Amyotrophic lateral sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Success rate of weaning from mechanical ventilation in both groups | 48 Hours after weaning
  (The trial will be considered a successful weaning trial if the patient passed 48 hours without the need for neither invasive nor non-invasive ventilation)

SECONDARY OUTCOMES:
• Rapid shallow breathing index (RSBI) and its correlation with ultrasound derived variables | baseline
• Days of ventilation (before weaning trial) in correlation to diaphragmatic dysfunction | baseline
• Number of weaning trials prior to inclusion in the study | baseline

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mohamed moukhtar, MD, Principal Investigator — professor of anesthesiology cairo university; waleed ibrahim Hamimmy, MD, Principal Investigator — professor of anesthesiology cairo university; akram shahat Eladawy, MD, Principal Investigator — assistant professor of anesthesiology cairo university; ahmed muhamed lotfy, MD, Principal Investigator — lecturer of anesthesiology cairo university; mina adolf helmy, MSc, Principal Investigator — assistant lecturer of anesthesiology cairo university
Locations (1):
- Cairo University-Manial, Cairo, Egypt

REFERENCES:
- [Background] El-Khatib MF, Bou-Khalil P. Clinical review: liberation from mechanical ventilation. Crit Care. 2008;12(4):221. doi: 10.1186/cc6959. Epub 2008 Aug 6. PMID 18710593
- [Background] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Background] Fagon JY, Chastre J, Hance AJ, Montravers P, Novara A, Gibert C. Nosocomial pneumonia in ventilated patients: a cohort study evaluating attributable mortality and hospital stay. Am J Med. 1993 Mar;94(3):281-8. doi: 10.1016/0002-9343(93)90060-3. PMID 8452152
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Heunks LM, van der Hoeven JG. Clinical review: the ABC of weaning failure--a structured approach. Crit Care. 2010;14(6):245. doi: 10.1186/cc9296. Epub 2010 Dec 8. PMID 21143773
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Background] Jiang JR, Tsai TH, Jerng JS, Yu CJ, Wu HD, Yang PC. Ultrasonographic evaluation of liver/spleen movements and extubation outcome. Chest. 2004 Jul;126(1):179-85. doi: 10.1378/chest.126.1.179. PMID 15249460